CLINICAL TRIAL: NCT03716622
Title: A Comparison of Clarithromycin-based and Furazolidone-based Bismuth-containing Regimens for H. Pylori Eradication
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, director of Qilu Hospital gastroenterology department, Shandong University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2018SDU-QILU-G112
Record Dates: First submitted 2018-10-21; First posted 2018-10-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Helicobacter Pylori
Keywords: Helicobacter Pylori; furazolidone; clarithromycin; bismuth-containing quadruple regimen
MeSH Terms: interventions — Furazolidone; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bismuth-clarithromycin-containing group (Active Comparator): Patients in bismuth-clarithromycin-containing group will receive lansoprazole (Takepron) 30mg po bid, amoxicillin 1000mg po bid, bismuth subcitrate (Colloidal Bismuth Pectin) 200mg po bid, and clarithromycin (Klacid) 500mg po bid for 14d
  Interventions: Drug: Clarithromycin
- bismuth-furazolidone-containing quadruple group (Experimental): patients in bismuth-furazolidone-containing quadruple group will receive lansoprazole (Takepron) 30mg po bid, amoxicillin 1000mg po bid, bismuth subcitrate (Colloidal Bismuth Pectin) 240mg po bid, and furazolidone (Liteling) 100mg po bid for 14d
  Interventions: Drug: Furazolidone

INTERVENTIONS:
Drug: Furazolidone — bismuth-furazolidone-containing quadruple regimens
  Arms: bismuth-furazolidone-containing quadruple group
Drug: Clarithromycin — bismuth-clarithromycin-containing quadruple regimens
  Arms: bismuth-clarithromycin-containing group

SUMMARY:
We aim to assess and compare the effectiveness of clarithromycin- and furazolidone-based regimens as primary therapies in eradicating H. pylori.

DETAILED DESCRIPTION:
Helicobacter pylori plays a pivotal role in many diseases such as peptic ulcer disease and MALT lymphomas. And the prevalence of H. pylori is increasing in some parts of the world.

However, the eradication becomes increasingly difficult due to the growing antibiotic resistance. Bismuth-containing quadruple regimens are now recommended to serve as first-line therapies. Bismuth-clarithromycin-containing and bismuth-furazolidone-containing quadruple regimens are both in the list of the first regimens. And recent antimicrobial susceptibility tests showed us that the clarithromycin was increasingly resisted while furazolidone remained hardly resisted. The comparison between the effects of bismuth-clarithromycin-containing and bismuth-furazolidone-containing quadruple regimens is not so clear.

ELIGIBILITY:
Inclusion Criteria:

* Patients, aged between 18 and 75years old, with positive H. pylori infection that was not eradicated by previous therapies are included. The H. pylori infection is confirmed by the positive rapid urease test or 13C-breath test.

Exclusion Criteria:

* Patients with significant underlying disease including liver, cardiac, pulmonary, and renal diseases, neoplasia, coagulopathy and genetic diseases, history of gastric surgery, pregnancy, breast-feeding, active gastrointestinal bleeding, the use of PPI, NSAID or antibiotics during the 4 weeks prior to enrolment, and previous history of allergic reactions to any of the medications used in this protocol. Patients previously treated with H. pylori eradication regimens or those unwilling to participate in the study were also excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
the eradication rate of the two groups | 26 months

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zuo, MD,PhD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu hosipital, Jinan, Shandong, China